CLINICAL TRIAL: NCT05334914
Title: An Online/In Person Program Assessing Acceptance Commitment Therapy Matrix Plus Contingency Management for Methamphetamine Use Disorder in Women and Gender Non-Conforming Individuals
Brief Title: ACT for Methamphetamine Use Disorder in Women and Gender Non-Conforming Individuals
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Bernard Le Foll, Senior Scientist, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMH CCI ACT
Record Dates: First submitted 2022-04-07; First posted 2022-04-19 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Methamphetamine Abuse; Methamphetamine-dependence
Keywords: Methamphetamine use disorder; Acceptance commitment therapy; Contingency management; Motivational interviewing; App-based interventions; Telehealth; Women; Gender Non-Conforming; Non-binary
MeSH Terms: interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: Single-arm, open-label, feasibility trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Other): Participants will complete the baseline session, a 1:1 motivation building session, and 8 weeks of ACT group therapy. They will then complete a final study visit and a follow-up study visit to occur 6 month after the end of therapy.
  Interventions: Behavioral: Acceptance Commitment Therapy

INTERVENTIONS:
Behavioral: Acceptance Commitment Therapy — ACT: Consists of 15 sessions, twice per week. Each session is approximately 2.5 hours including breaks. Clients cover 3 modules (OPEN, ACTIVE, AWARE). Any participant who requires access to a device for any part of the study will be provided with one for the duration of the study.
  CM: Participants will be given progressive compensation for session attendance via gift cards or e-gift cards amounting to $520.
  Motivation Building Session: The study clinician will meet with each of the participants to explain the process of the therapy, reinforce expectations, and address any concerns or hesitations, and build motivation and commitment to fully engage in the program.
  ChillTime App Participants rate their emotional state and choose a coping strategy (either physical, emotional, cognitive or spiritual). The app's algorithm learns the individual's strategy preferences over time, allowing for more personalized suggestions. Participants are also able to access coping strategies ad hoc.
  Other Names: Contingency Management; Motivation Building; App-Based Therapy

SUMMARY:
This study aims to assess the feasibility, acceptability and preliminary effectiveness of Acceptance Commitment Therapy, in conjunction with motivation enhancement, and the use of the ChillTime App, in reducing methamphetamine use in women with MUD with or without co-occurring psychiatric disorders. This intervention is designed to be delivered remotely (e.g., participants can complete the entire study from home), with the option for in person attendance if it is not feasible or safe for participants to attend from home.

DETAILED DESCRIPTION:
Women and gender non-conforming (GNC) individuals with methamphetamine use disorder (MUD) are a particularly vulnerable population in need of complex interventions that can address the range of severe clinical issues with which they often present. However, there are currently no existing psychosocial interventions that are considered preferred for MUD generally, much less in women and GNC individuals with complex psychological profiles and social positioning.

Complex interventions refer to a multifaceted approach to the treatment of psychiatric conditions and may consist of several therapeutic modalities (e.g., behavioural, pharmacological, technological, family engagement; May et al., 2007). These interventions are designed with the intent that they are easy to incorporate into everyday clinical practice (May et al., 2007) and will be effective in treating members of the general population, who present with complex conditions.

As such, the investigators aim to assess the feasibility, acceptability, and effectiveness of a) Acceptance Commitment Therapy delivered in a group format twice weekly, b) an intrinsic motivation building session and contingency management (i.e., progressive monetary incentivizing) targeting session attendance, and c) the ChillTime App to promote the use of emotional coping strategies between sessions.

The program will be 15 sessions/8 weeks long with outcome data collected at a 1-month follow up to assess longevity of effects on MUD harm reduction, abstinence, and mental health.

The investigators will recruit 60 participants through existing service providers in the Greater Toronto Area. As a broader aim of our study is to promote generalizability to the community and ensure the intervention will be accessible to all women and GNC individuals with MUDs, the following are implemented: a) group sessions will be delivered remotely, with an option for in person attendance if remote access is not feasible; b) broad inclusion criteria (e.g., not excluding on the basis of other mental health/substance use comorbidities); and c) qualitative interviews during which patient perspectives will be gathered and the intervention will be adapted accordingly, where warranted. Results will be used to inform a large-scale, randomized, controlled clinical trial.

Study Design: Each participant will undergo a screening/baseline assessment where they will complete clinical assessments to determine eligibility. Following the screening period and signing of the consent form, the study clinician will schedule a 1:1 motivation building session with participants. Participants will be given the 8-week ACT group schedule and research staff will assist them with downloading the ChillTime App. Over the course of the 8-week treatment, participants will learn coping and emotional regulation strategies, and will be able to access additional strategies through the use of the app. After the last group session, participants will once again complete clinical and quality of life assessments. The research staff administering the adverse events and outcome measures will not be the study clinician. The same questionnaires will be used at the 1 month follow-up, along with a qualitative interview asking about their satisfaction with and experience in the program as well as any changes in drug use reflective of harm reduction (e.g., stopped sharing pipes). Participants who missed a session will be offered the chance to make it up 1-1 with the study therapist; participants who dropped out of the group will also be contacted for an Early Termination Visit and will be asked to identify their reasons for dropping out.

ELIGIBILITY:
Inclusion Criteria:

* Meet SCID DSM-5 criteria for Methamphetamine Use Disorder
* Over the age of 18
* Female, woman, or non-binary and comfortable participating in women's group
* Capacity to provide informed consent
* Adequate English language abilities

Exclusion Criteria:

* Experiencing acute or unmedicated psychosis that would reasonably prevent them from engaging in and/or benefiting from the intervention
* Experiencing acute and severe suicidal ideation such that institutionalization and supervised care is warranted
* Experiencing severe cognitive deficits that would reasonably prevent them from consenting, engaging in, and/or benefiting from the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Identifies as female, woman, or non-binary and is comfortable participating in a women's group
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of intervention | Immediately after intervention
  Rates of eligible participants who agree to participate in the study intervention; Rates of retention in program (e.g., number of participants that completed all 15 sessions, number of participants that completed at least a full dose of 10 sessions, number of participants that dropped out before 10 sessions); Rate of use of ChillTime App
Acceptability of intervention | 1 month follow-up
  Acceptance and understanding of the program using qualitative assessments at the end of study and the Client Satisfaction Questionnaire

SECONDARY OUTCOMES:
Changes in methamphetamine use via the timeline followback (TLFB) | Baseline, immediately after intervention, 1 month follow-up
  The Timeline Followback (TLFB) is a method that can be used as a clinical and research tool to obtain a variety of quantitative estimates of methamphetamine use over the past 7-days
Changes in methamphetamine use via urinalysis | Baseline, immediately after intervention, 1 month follow-up
  Liquid chromatography/mass spectrometry will be used to provide qualitative (yes/no) assessments of presence of methamphetamine in urine
Changes in other substance use via the Timeline Followback (TLFB) | Baseline, immediately after intervention, 1 month follow-up
  The Timeline Followback (TLFB) is a method that can be used as a clinical and research tool to obtain a variety of quantitative estimates of other drug use over the past 7-days
Changes in anxiety via the Generalized Anxiety Disorder-7 (GAD-7) | Baseline, immediately after intervention, 1 month follow-up
  The Generalized Anxiety Disorder Assessment (GAD-7) is a seven-item instrument that is used to measure or assess the severity of generalised anxiety disorder (GAD). Each item asks the individual to rate the severity of his or her symptoms over the past two weeks.
Changes in depression via the Patient Health Questionnaire-9 (PHQ-9) | Baseline, immediately after intervention, 1 month follow-up
  The PHQ-9 is the nine item depression scale of the patient health questionnaire. The nine items of the PHQ-9 are based directly on the nine diagnostic criteria for major depressive disorder in the DSM-IV. The PHQ-9 can function as a screening tool, an aid in diagnosis, and as a symptom tracking tool that can help track a patient's overall depression severity as well as track the improvement of specific symptoms with treatment.
Changes in trauma symptoms via the Trauma Screening Questionnaire (TSQ) | Baseline, immediately after intervention, 1 month follow-up
  The TSQ is a 10-item symptom screen that was designed for use with survivors of all types of traumatic stress. The TSQ is based on items from the PTSD Symptom Scale - Self Report (PSS-SR; Foa et al., 1993) and has five re-experiencing items and five arousal items.
Changes in acceptance commitment skills via the Acceptance and Action Questionnaire [AAQ-2 | Baseline, immediately after intervention, 1 month follow-up
  This 4-item measure uses 0-4 scale (0 = Not at All True; 4 = Very True) with lower sores correlating with higher psychological flexibility.
Changes in cravings/urges for methamphetamine via the Brief Substance Craving Scale BSCS | Baseline, immediately after intervention, 1 month follow-up
  The BSCS is a 16 item, self-report instrument assesses craving for cocaine and other substances of abuse over a 24 hour period. Intensity and frequency of craving are recorded on a five-point Likert scale
Changes in quality of life, including well-being, relationships, social activities, personal fulfillment and recreation via the World Health Organization Quality of Life- BREF [WHOQOL-BREF] | Baseline, immediately after intervention, 1 month follow-up
  Measures Quality of Life defined as an individual's perception of their position in life in the context of the culture and value systems in which they live and in relation to their goals, expectations, standards and concerns.
Drug use or harm reduction practices at the end of the study via semi-structured interviews | 1 month follow up
  Semi-structured interview with member of research team
Barriers to engaging in the intervention using qualitative assessments at the end of study | 1 month follow up
  Semi-structured interview with member of research team
Engagement in treatment | Immediately after intervention
  The Treatment Engagement Rating Scale was developed to assess patient engagement and behaviour change after an 8 week intervention; and will be adapted for this population. It is filled out by the study clinician for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Le Foll, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No